CLINICAL TRIAL: NCT02819817
Title: A Parallel Group Double Blind Placebo Randomised Controlled Trial (RCT) of Topical Aloe Vera Gel in Emergency Department (ED) Patients Presenting With Simple Traumatic Wounds
Brief Title: A Trial of Topical Aloe Vera Gel in Emergency Department Patients Presenting With Simple Traumatic Wounds
Acronym: ALOE
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: MHRA CTA rejected due to no UK MHRA MA certificate or equivalent product info
Sponsor: NHS Lothian (Other Government)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC16063
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Injuries and Wounds
Keywords: Aloe Vera, wound, healing
MeSH Terms: conditions — Wounds and Injuries | interventions — Aloe vera gel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aloe Vera Gel (Experimental): Experimental gel placed in identical opaque tube as placebo gel.
  Interventions: Drug: Aloe Vera Gel
- Ultrasound Gel (Placebo Comparator): Placebo placed in identical opaque tube as experimental gel.
  Interventions: Other: Ultrasound gel
- Standard care (No Intervention): Standard care

INTERVENTIONS:
Drug: Aloe Vera Gel — The participant will be asked to place the allocated substance onto the wound twice daily and cover with a supplied dressing on each occasion for 1 week.
  Other Names: Aloe Vera Gel (LIFEPLAN)
  Arms: Aloe Vera Gel
Other: Ultrasound gel — The participant will be asked to place the allocated substance onto the wound twice daily and cover with a supplied dressing on each occasion for 1 week.
  Other Names: Sterile (AQUASONIC 100) ultrasound transmission gel
  Arms: Ultrasound Gel

SUMMARY:
This is a double blind placebo-controlled RCT comparing the speed of healing of simple traumatic wounds with Aloe Vera gel compared to both control (Ultrasound gel) and standard care.

DETAILED DESCRIPTION:
Simple traumatic wounds are a common presenting symptom to the ED affecting thousands of patients worldwide every day. Aloe Vera is a natural product that has been linked to better healing both anecdotally and in animal studies. A recent Cochrane review failed to find any human studies on acute wounds such as those seen in the ED. The aim of this study is to see whether Aloe Vera gel improves the wound healing time in these patients. We plan to enrol 270 participants presenting to the Royal Infirmary of Edinburgh ED with simple traumatic wounds into a randomised controlled trial. Participants will be assessed at baseline using the Bates-Jensen wound assessment tool. They will be then be randomized to one of three groups, and allocated to receive either Aloe Vera gel, control (Ultrasound gel) or standard care. The participants in the two gel groups will have identical packaging and the treating clinician will be unaware as to which group they are allocated. They will be asked to place the allocated substance onto the wound twice daily and cover with a supplied dressing on each occasion for 1 week. All groups will be asked to return to the ED for a repeat Bates-Jensen wound assessment, and will also be asked to record the number of days that their wound took to heal. The gel groups will have assessment of product usage. Participants will also be telephoned at 3 weeks. Primary outcome will be number of days for wound to heal. Secondary outcome will be change in Bates-Jensen wound assessment score between baseline and day 10, change in wound size between baseline and day 10 and baseline and day 21, changes in wound characteristics at day 21 as reported by participants, wound infection rate, participant satisfaction and participant compliance with treatment.

ELIGIBILITY:
Inclusion Criteria: Patients deemed by their treating clinician to have a simple traumatic wound will be considered for enrolment.

Exclusion Criteria:

1. Known allergy to either Aloe Vera or ultrasound gel
2. Patients under 16 year of age
3. No telephone number for follow-up
4. Patient lacking capacity
5. Patient currently using antibiotics
6. Patient having a puncture or bite wound
7. Patient having underlying tendon or bone involvement or wound overlying a joint
8. Patients with burn wounds
9. Wounds more than 24 hours old
10. Patient unable/unwilling to attend follow-up
11. Patients unable to self administer treatment.
12. Wound that treating clinician would not routinely dress e.g. facial wounds (face, ear, eyebrow, nose, lip, eyelid, scalp), mucosa and hair covered areas, or wounds that require specialist dressing
13. Self reported pregnancy
14. Patients with a known allergy to the study dressing
15. Patients currently recruited in another clinical trial
16. Patients already recruited in the ALOE Study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Number of days for wound to heal (defined as epithelial closure without discharge or scab formation) | Day 21 (+/- 2 days)

SECONDARY OUTCOMES:
Numerical change in Bates-Jensen wound assessment score between baseline and day 10 (+/- 2 days) | Baseline and day 10 (+/- 2 days)
Size (width and height in mm) of wound at baseline, day 10 (+/- 2 days), and day 21 (+/- 2 days) | Baseline, day 10 (+/- 2 days) and day 21 (+/- 2 days)
Characteristics (visibility of wound edges and leakage from wound) as reported by participant at day 21 (+/- 2 days) | Day 21 (+/- 2 days)
Wound infection rate | Day 21 (+/- 2 days)
Participant satisfaction score | Day 21 (+/- 2 days)
Participant treatment compliance (i.e. the total weight of gel used) | Day 10 (+/- 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Reed, MA FRCEM MD, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No